CLINICAL TRIAL: NCT05078151
Title: A Study to Clinically Qualify Whole-Body Diffusion-Weighted Magnetic Resonance Imaging (MRI) in Patients With Metastatic Castration Resistant Prostate Carcinoma With Bone Metastases
Brief Title: Whole-Body Diffusion-Weighted Magnetic Resonance Imaging (MRI) as a Response Biomarker for Metastatic Prostate Cancer
Acronym: iPROMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Collaborators: Prostate Cancer Foundation (Other); Instituto de Salud Carlos III (Other Government); Hospital Vall d'Hebron (Other); Fundacio Puigvert (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ipromet21
Record Dates: First submitted 2021-09-28; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer Metastatic
Keywords: response biomarker; functional imaging; MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic prostate cancer (Other): Patients will receive whole-body MRI with diffusion-weighted imaging at baseline and after 4 and 8 weeks of treatment.
  Interventions: Diagnostic Test: Whole-Body Diffusion Weighted MRI

INTERVENTIONS:
Diagnostic Test: Whole-Body Diffusion Weighted MRI — MRI at baseline, after four and eight weeks of treatment and at disease progression or treatment discontinuation.

SUMMARY:
The skeleton is the most frequent organ of distal metastases in prostate cancer, often representing the only site of metastatic disease. Still, assessment of response and progression to therapies in bone metastases remains a major unmet need, to aid treatment switch decisions, detecting primary/secondary resistance and to optimize drug development. The currently used standard imaging techniques, computed tomography (CT) and bone scintigraphy (BS), do not depict the true extent of bone metastases and are suboptimal in capturing biological changes occurring in response to treatment.

This results in treatment switch decisions too often being based on PSA changes, which is neither a surrogate of survival, nor an optimal response biomarker.Diffusion-weighted imaging (DWI) is a functional magnetic resonance imaging (MRI) technique that studies the movement of water molecules within a tissue and provides valuable information about the tissue microstructure and cellularity. Whole body MRI with DWI is highly accurate for bone metastases detection, outperforming the standard CT and BS and other imaging techniques when assessing bone metastases.

The investigators hypothesise that DWI changes are a response biomarker in bone metastases from metastatic castration resistant prostate cancer (mCRPC); these DWI changes can be detected as early as after 4 weeks of systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 or over years old.
* Patients with castration resistant prostate cancer.
* Evidence of bone metastases by any imaging technique.
* Patients due to start treatment with abiraterone or enzalutamide. In the exploratory cohorts, we will include patients due to start treatment with other systemic therapies for advanced prostate cancer (A-taxanes, B-radiopharmaceuticals, C-other therapies).
* Written (signed and dated) informed consent.

Exclusion Criteria:

* Contraindications to MRI.
* Inability of patient to tolerate whole body MRI (e.g. claustrophobia).
* Patients who have received radiotherapy within the last three months and with no bone metastases outside the radiotherapy field.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in diffusion-weighted MRI as response biomarker | 8 weeks after treatment
  Apparent Diffusion Coefficient (ADC) percentage change in responders vs non-responders to systemic treatment in patients with CRPC and bone metastases

SECONDARY OUTCOMES:
Early response biomarker identification | 4 weeks after treatment
  Apparent Diffusion Coefficient (ADC) percentage change in responders vs non-responders to systemic treatment in patients with CRPC and bone metastases
Intra-tumor heterogenous response evaluation | 4 and 8 weeks after treatment and at disease progression by standard criteria, on average 1 year
  To use diffusion-weighted MRI for identifying anatomic regions of subclonal resistance to systemic treatment and study tumour evolution.

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron Institute of Oncology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No